CLINICAL TRIAL: NCT07015463
Title: Evaluation of a Health Literacy Intervention on Patients Suffering From Hypertension in Primary Care
Acronym: IHTALi
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2023/53
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Hypertension
Keywords: health literacy; intervention; high blood pressure
MeSH Terms: conditions — Hypertension | interventions — Health Literacy

STUDY DESIGN:
Intervention Model Description: mixed-method cluster randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General Practitioner (GP) exposed to the intervention (Experimental): The intervention will be developed during the first phase according to the theoretical conceptual model Health proposed by Bas Geboers. The final intervention will take the form of a standardized intervention guide containing the elements of the intervention.
  Five targets respond to the theoretical model:
  * Healthcare professionals, through interventions enabling them to improve their skills regarding health literacy (HL) (such as identifying HL problems in their patients, increasing their communication skills, etc.)..
  * The patient and their entourage, through interventions that strengthen the support of their entourage (family, peers, etc.).
  * Patients, through empowerment interventions.
  * Patient-health system interaction, through interventions aimed at improving communication between patients and healthcare professionals.
  * Improving blood pressure control access, through interventions focused on reducing access barriers or policies to improve the quality of care.
  Interventions: Other: Multi-component intervention in health literacy
- GP of the control group (No Intervention): GP following usual guidelines

INTERVENTIONS:
Other: Multi-component intervention in health literacy — Multi-component intervention aiming at increasing the health literacy of patients suffering from hypertension, in achieving the target blood pressure goal three months after the start of the intervention in poorly controlled hypertensive patients
  Arms: General Practitioner (GP) exposed to the intervention

SUMMARY:
Hypertension affects 30% of the French population, but only 25% of hypertensive patients meet therapeutic targets, largely due to a limited adherence to lifestyle and medication guidelines (34%). Improving adherence is crucial to better blood pressure control and preventing complications. Health literacy (HL), defined by Sørensen as the ability to access, evaluate, and use health information for decision-making, has been proved associated with better adherence. Various tools, such as the "Teach-Back" method, can enhance HL but are underutilized in France due to lack of awareness and training. The objective of this study is to evaluate the effectiveness of a multi-component intervention aimed at increasing the health literacy of patients suffering from hypertension, in achieving the target blood pressure goal three months after the start of the intervention in poorly controlled hypertensive patients. The intervention will include tools (such as communication techniques) enabling physicians to enhance the health literacy of their patients.

DETAILED DESCRIPTION:
The study comprises two phases. The first phase will involve a qualitative analysis, during which semi-structured interviews will be conducted to understand the constraints, expectations, and needs of both physicians and patients for the intervention. After this phase, an intervention following the Health Literacy Intervention Model will be constructed, through a consensus method .

The second phase of the study will be a mixed-method evaluation of the intervention's effectiveness. Initially, a cluster-randomized trial will be conducted. Thirty-six physicians will participate and randomized into either the control group or the intervention group. Each physician will recruit approximately 5 patients. Patients will undergo a pre-inclusion visit, an inclusion visit, and then three follow-up visits (at 3 and 6 months). Finally, all participating physicians and a subsample of 30 patients will take part in the qualitative study to assess the perceived effectiveness of the intervention.

ELIGIBILITY:
Inclusion criteria:

Phase 1: Co-construction of the Intervention

o In this phase, physicians and patient representatives from patient associations or recruited through physicians will be enrolled.

Phase 2: Evaluation of the Intervention's Effectiveness

Inclusion Criteria for Investigating Physicians

General practitioners practicing:

* In individual offices, in non-multidisciplinary group practices
* Or in multidisciplinary health centers or health centers
* In Nice, Bordeaux, and Lille
* Who have expressed their non-opposition
* Willing to participate in the qualitative evaluation

Inclusion Criteria for Patients

* Adult French-speaking patients, able to read and write
* Suffering from essential uncontrolled and treated hypertension treated measured by home self-monitoring
* Owning a mobile phone (to be contacted for the study and to receive reminder by phone)
* Able to self-measure his/her blood pressure at home
* Who have expressed their non-opposition

Inclusion for qualitative interviews Only individuals from the intervention group will be asked to participate in these interviews.

* All physicians who recruited patients for the trial will be invited to participate.
* A subsample of 30 patients (10 per city), selected according to the principle of maximum variation (ensuring diversity in age and gender)

Exclusion criteria:

Phase 1: Co-construction of the intervention

No exclusion criteria will be applied for this phase.

Phase 2: Evaluation of the effectiveness of the intervention

Exclusion Criteria for Investigating Physicians

* GP who participated in the first phase of co-construction.
* GP from a health center where a collaborator has already been recruited for the study.
* GP working in collaboration with an Asalée nurse.

Exclusion Criteria for Patients

* Patient suffering from secondary hypertension.
* Patient with severe cognitive impairment or dementia.
* Patients already performing regular self-monitoring of their blood pressure.
* Healthcare professionals.
* Patient under legal protection, guardianship, or curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 255 (Estimated)
Dates: Start 2025-07-31 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with a home-measured blood pressure within the therapeutic target | three months after the implementation of the intervention
  Proportion of patients with a home-measured blood pressure within the therapeutic target three months after the implementation of the intervention (systolic blood pressure below 140 mm Hg for patients under 80 years old or below 150 mm Hg for patients 80 years and older).

SECONDARY OUTCOMES:
Improvement in achieving the target blood pressure six months after the start of the intervention | six months after the intervention
  Proportion of patients with blood pressure,within the therapeutic target (defined as systolic blood pressure <140 mmHg for patients under 80 years old, or <150 mmHg for patients aged 80 and over), in both groups (intervention vs. control).
Improvement in achieving the target blood pressure at three months after the start of the intervention, in GPs | Three months after the intervention
  Proportion of patients with blood pressure within the therapeutic target of the intervention (defined as systolic blood pressure <140 mmHg for patients under 80 years old, or <150 mmHg for patients aged 80 and over), in both groups (intervention vs. control), measured in general practitioners' offices on the day of the follow-up visit.
Improvement in achieving the target blood pressure at six months after the start of the intervention, in GPs | Six months after the intervention
  Proportion of patients with blood pressure within the therapeutic target of the intervention (defined as systolic blood pressure <140 mmHg for patients under 80 years old, or <150 mmHg for patients aged 80 and over), in both groups (intervention vs. control), measured in general practitioners' offices on the day of the follow-up visit.
Health Literacy Level | 6 months after the intervention
  Patients' health literacy level regarding hypertension measured by the score obtained on the HLS-EU16
Adherence to treatment scale using Girerd questionnaire | Baseline, three and six months
  Adherence will be assessed by an investigator over the phone
Effect of the Intervention by Social Categories | Baseline, three and six months
  The proportion of patients with blood pressure within the therapeutic target will be assessed in relation to an individual index of social disadvantage (EPICES score and income level measured at baseline). The proportion of patients achieving the target blood pressure will be described by EPICES score quintiles and income level categories at each of the three time points.
Effective adoption of tools in the intervention group | At the end of the follow-up, for each patient
  Frequency of use of the recommended tools for each patient, and eventually extended use for other conditions
Perceived effectiveness by patients | During the six months after the end of the trial
  Patients' appropriation of the intervention and its impact on health-promoting behaviors, their experience and perceptions in managing the disease, and the evolution of their representations regarding their care.
Perceived effectiveness from the perspective of healthcare professionals | During the six months after the end of the trial
  Actual implementation of the intervention by professionals in the intervention group. And professionals' perceived appropriation of the intervention and its impact on professional and organizational practices
Choose and adapt tools of intervention to the context of primary care | Before the beginning of the randomized trial
  Proposition of a theory-based intervention using qualitative interviews. A standardized intervention based on the Health Literacy Intervention Model, developed in collaboration with physicians and hypertensive patients, which can be easily integrated into general practitioners' practices will be developped.
Investigate the factors influencing the acceptability and effectiveness of the LS intervention | Before the beginning of the randomized trial
  Understanding of implementation contexts/ Usual behaviors of healthcare professionals/Difficulties encountered in practice and with existing health literacy tools/Needs and expectations regarding the intervention, as expressed by patient representatives and physicians (working in general practices or multidisciplinary health centers)

CONTACTS AND LOCATIONS:
Overall Officials: Florence FRANCIS-OLIVIERO, MD, Principal Investigator — IRDES

IPD SHARING:
Plan to Share IPD: No